CLINICAL TRIAL: NCT01588470
Title: Myocardial Dysfunction in Type 2 Diabetes Mellitus (T2DM) - Role of Intramyocellular Lipid Content and Mitochondrial Dysfunction in Myocardial Insulin Resistance and Their Correction With Pioglitazone
Brief Title: Myocardial Dysfunction in Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Ralph DeFronzo, Professor & Division Chief, Department of Medicine, Division of Diabetes, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM20060280; T001 (Other Grant/Funding Number: Takeda)
Record Dates: First submitted 2012-03-19; First posted 2012-05-01 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes; Coronary Heart Disease
Keywords: diastolic function; mitochondria; pioglitazone; pericardial fat
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Disease | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: this study includes single arm intervention with pioglitazone. T2DM individuals will be studied at baseline and after 6 months treatment.
  as a reference group, healthy subjects will be studied in cross sectional fashion. Because healthy subjects will not be treated nor restudied at 6 months, they can not be considered a separate arm in the study but rather a reference group
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pioglitazone (Experimental): Only subjects with T2DM or non-diabetic subjects with coronary heart disease will receive Pioglitazone
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: pioglitazone — 45 mg per day for 6 months
  Other Names: Actos

SUMMARY:
The purpose of this study is to examine the existence of heart abnormalities in patients with diabetes and the effect of pioglitazone in correcting these abnormalities.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES

1. To quantitate myocardial insulin sensitivity using positron emission tomography (PET) with 18F-deoxyglucose in type 2 diabetes mellitus (T2DM) and control subjects.
2. To quantitate pericardial fat using magnetic resonance spectroscopy in T2DM and control subjects.
3. To quantitate cardiac function using magnetic resonance imaging and echocardiography in T2DM and control subjects.
4. To examine the effect of pioglitazone on myocardial insulin sensitivity, pericardial fat content, and cardiac function.

SECONDARY OBJECTIVES To examine the relationships between myocardial insulin sensitivity, pericardial fat content, and cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
* Patients may be of either sex. Female patients must be non-lactating and must either be at least one year post-menopausal, or be using adequate contraceptive precautions (i.e. oral contraceptives, approved hormonal implant, intrauterine device, diaphragm with spermicide, condom with spermicide), or be surgically sterilized (i.e. bilateral tubal ligation, bilateral oophorectomy). Female patients who have undergone a hysterectomy are eligible for participation in the study. Female patients (except for those patients who have undergone a hysterectomy or a bilateral oophorectomy) are eligible only if they have a negative pregnancy test throughout the study period
* Patients must range in age from 18 to 75 years, inclusive.
* Patients with type 2 diabetes must be drug naïve, receiving monotherapy with metformin or with a sulfonylurea, or combination therapy with both: metformin & sulfonylurea.
* Patients must have the following laboratory values:

  * Hematocrit ≥ 34 vol%
  * Serum creatinine ≤ 1.8 mg/dl
  * AST (SGOT) ≤ 2.5 times upper limit of normal
  * ALT (SGPT) ≤ 2.5 times upper limit of normal
  * Alkaline phosphatase ≤ 2 times upper limit of normal
* Patients must have been on a stable dose of allowed chronic medications for 30 days prior to entering the study.
* Only subjects whose body weight has been stable (±3-4 pounds) over the three months prior to study will be included.

Exclusion Criteria:

* Patients must not have type 1 diabetes.
* Patients must not be receiving any medications with known adverse effects on glucose tolerance (except metformin or a sulfonylurea) unless the patient has been on stable doses of such agents for the past three months before entry into the study. Patients may be taking stable doses of estrogens or other hormonal replacement therapy, if the patient has been on these agents for the prior three months. Patients taking systemic glucocorticoids are excluded.
* Patients with a history of clinically significant heart disease (New York Heart Classification greater than class 2; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
* Patients with hematocrit < 34% will be excluded.
* Patient who were exposed to any procedure involves radiation exposure and his total radiation dose equivalent exceeds 5 rem during the past year will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A DeFronzo, MD, Principal Investigator — University of Texas

IPD SHARING:
Plan to Share IPD: No
IPD data will not be available for other researchers. However, a manuscript describing the study results is under review for publication in the medical literature

REFERENCES:
- [Derived] Clarke GD, Solis-Herrera C, Molina-Wilkins M, Martinez S, Merovci A, Cersosimo E, Chilton RJ, Iozzo P, Gastaldelli A, Abdul-Ghani M, DeFronzo RA. Pioglitazone Improves Left Ventricular Diastolic Function in Subjects With Diabetes. Diabetes Care. 2017 Nov;40(11):1530-1536. doi: 10.2337/dc17-0078. Epub 2017 Aug 28. PMID 28847910

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone: Only subjects with T2DM or non-diabetic subjects with coronary heart disease will receive Pioglitazone
  pioglitazone : 45 mg per day for 6 months
Period: Overall Study
Arm/Group | Pioglitazone
Started | 130 (First enrolled April 2007)
Completed | 50 (Completed Dec. 2011)
Not Completed | 80

BASELINE CHARACTERISTICS:
Arm/Group | Pioglitazone
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in E to A Ratio
Description: The E to A ratio is a marker of the function of the left ventricle of the heart. It represents the ratio of peak velocity flow in early diastole (the E wave) to peak velocity flow in late diastole caused by the atrial contraction (the A wave) This is measured using ultrasound-based cardiac imaging. In a healthy heart the E velocity is greater than the A velocity.
Time Frame: Baseline and 6-months Post Treatment
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Baseline: Measure of E to A Ratio to determine which subjects will receive
  pioglitazone: 45 mg per day for 6 months
- E to A Ratio After Pioglitazone Treatment: Only subjects with T2DM or non-diabetic subjects with coronary heart disease will receive Pioglitazone
  pioglitazone: 45 mg per day for 6 months
Arm/Group | Baseline | E to A Ratio After Pioglitazone Treatment
Number analyzed (Participants) | 130 | 50
Ratio | 1.04 (0.28) | 1.25 (0.38)
Statistical Analysis 1: Comparison: E to A Ratio After Pioglitazone Treatment; Test type: Superiority; p < 0.01, ANOVA

2. Primary Outcome: Myocardial Glucose Uptake
Description: Measurement of change in myocardial glucose uptake from baseline to 6 months of treatment with pitoglitazone
Time Frame: Baseline and 6-months Post Treatment
Population: Study participants who met eligibility criteria
Measure: Mean (Standard Deviation); unit: uM/min/g
Groups:
- Baseline: Only subjects with T2DM or non-diabetic subjects with coronary heart disease measurement of Myocardial Glucose Uptake (MGU) at before Pioglitazone administration.
- Pioglitazone: Subjects with T2DM or non-diabetic subjects with coronary heart disease who received Pioglitazone -45 mg per day for 6 months
Arm/Group | Baseline | Pioglitazone
Number analyzed (Participants) | 130 | 24
uM/min/g | 0.24 (0.14) | 0.42 (0.13)

3. Secondary Outcome: Change in Hemoglobin A1c
Description: Change in hemoglobin A1c levels measured at 6 months
Time Frame: Baseline and 6-months Post Treatment
Population: Enrolled subjects that meet eligibility criteria as type 2 diabetics or non diabetic subjects with coronary heart disease
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Baseline; Pioglitazone: Only subjects with T2DM or non-diabetic subjects with coronary heart disease will receive Pioglitazone
  pioglitazone: 45 mg per day for 6 months
Arm/Group | Baseline | Pioglitazone
Number analyzed (Participants) | 130 | 12
percent | 6.7 (1.3) | 5.6 (0.8)
Statistical Analysis 1: Comparison: Baseline vs Pioglitazone; Test type: Superiority; p < 0.05, ANOVA; Mean Difference (Final Values) = -1.1

ADVERSE EVENTS:
Time Frame: data were collected over 6 months period
Arm/Group | Pioglitazone
All-Cause Mortality (participants affected / at risk) | 0/130
Serious Adverse Events (participants affected / at risk) | 0/130
Other Adverse Events (participants affected / at risk) | 2/130
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=130)
Mild weight gain ~2kg with ankle edema (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No